CLINICAL TRIAL: NCT06004817
Title: Evaluation of Severity in Juvenile Dermatomyositis and Adult-onset Dermatomyositis: a National Multicentric Retrospective Study
Brief Title: Evaluation of Severity in Juvenile and Adult-onset Dermatomyositis
Acronym: JADE
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI150
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Juvenile dermatomyositis: Dermatomyositis before 18 years-old
  Interventions: Other: evaluation of clinical severity
- Adult-onset dermatomyositis: Dermatomyositis from 18 years-old
  Interventions: Other: evaluation of clinical severity

INTERVENTIONS:
Other: evaluation of clinical severity — evaluation of clinical severity

SUMMARY:
Dermatomyositis (DM) are rare and heterogeneous systemic autoimmune diseases, characterized by the association of muscle inflammation, skin inflammation and vasculopathy. DM concern both adults and children. DM can be life-threatening (interstitial lung disease, infectious complications) and responsible of significant functional disability (muscle weakness). Age of onset appear to be an independent prognostic factor. Juvenile-onset DM is characterized by a higher frequency of calcinosis, skin ulceration and digestive vasculitis. In adults, interstitial lung disease and cancer are more frequent with higher mortality. Data concerning the comparison of the initial severity between juvenile and adult-onset DM are limited.

The main objective is to compare global severity between juvenile DM and adult-onset DM at initial diagnosis.

Secondary objectives are:

* to compare organ-specific severity between juvenile DM and adult-onset DM at diagnosis.
* to compare damage during follow-up and at last follow-up between juvenile DM and adult-onset DM.
* to compare activity at the last follow-up between juvenile DM and adult-onset DM.
* to compare iatrogenic complications between juvenile DM and adult-onset DM.

ELIGIBILITY:
Inclusion Criteria:

* Patient with dermatomyositis according to 2017 American College of Rheumatology (ACR)/ European Alliance of Associations for Rheumatology (EULAR) classification

Exclusion Criteria:

* Patient with cancer-associated dermatomyositis (within 3 years before or after diagnosis of dermatomyositis)
* Patient with antisynthetase syndrome

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed in pediatric and adult units during January 2010 and December 2022
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
number of patients with global severity | baseline (J0)
  presence of at least one criteria among: severe muscle disease (Childhood Myositis Assessment Scale
  - CMAS - score < 15, and/or Manual Muscle Testing 8 - MMT8 - score < 30, and/or Medical Research Council - MRC - muscle testing < 3, and/or dysphagia and/or swallowing difficulties), symptomatic interstitial lung disease (ILD), digestive vasculitis (digestive bleeding and/or vasculitis on CT-scan), myocarditis on cardiac MRI, severe skin ulcerations, intensive care unit admission

SECONDARY OUTCOMES:
number of patients with muscular severity | baseline (J0)
  presence of at least one of the following criteria: CMAS score < 15, MMT8 score < 30, MRC muscle testing < 3, dysphagia, swallowing difficulties
number of patients with pulmonary severity | baseline (J0)
  presence of symptomatic ILD
number of patients with digestive severity | baseline (J0)
  presence of digestive vasculitis: digestive bleeding and/or vasculitis on CT-scan
number of patients with cutaneous severity | baseline (J0)
  presence of severe skin ulcerations
myositis damage index (MDI) score | 2 years of follow-up, at 5 years of follow-up and at last follow-up
  myositis damage index (MDI) extent of damage score: from 0 (better outcome) to 38 (worse outcome)
number of patients with remission at last follow-up | up to 10 years
  absence of disease activity without any immunosuppressive/immunomodulatory treatment for at least 2 years
number of patients with disease activity at last follow-up | up to 10 years
  presence of at least one of the following criteria: elevated creatinine kinase (CK) level and/or recent muscle testing deterioration and/or muscle inflammation on MRI, and/or skin manifestations and/or progressive ILD

CONTACTS AND LOCATIONS:
Overall Officials: Paul Decker, MD, Principal Investigator — CHU NANCY
Locations (1):
- Chu Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No